CLINICAL TRIAL: NCT05022771
Title: A Phase 1A, First in Human, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of PMG1015 in Healthy Volunteers
Brief Title: A First in Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of PMG1015
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmongene Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMG1015-AUS-101
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Single Ascending Doses Cohort 1a (Experimental): Subjects will receive either Dose level 1 of PMG1015 or Placebo
  Interventions: Drug: PMG1015 Dose 1; Drug: Placebo
- Single Ascending Doses Cohort 1b (Experimental): Subjects will receive either Dose level 2 of PMG1015 or Placebo
  Interventions: Drug: PMG1015 Dose 2; Drug: Placebo
- Single Ascending Doses Cohort 1c (Experimental): Subjects will receive either Dose level 3 of PMG1015 or Placebo
  Interventions: Drug: PMG1015 Dose 3; Drug: Placebo
- Single Ascending Doses Cohort 1d (Experimental): Subjects will receive either Dose level 4 of PMG1015 or Placebo
  Interventions: Drug: PMG1015 Dose 4; Drug: Placebo
- Single Ascending Doses Cohort 1e (Experimental): Subjects will receive either Dose level 5 of PMG1015 or Placebo
  Interventions: Drug: PMG1015 Dose 5; Drug: Placebo
- Single Ascending Doses Cohort 1f (Experimental): Subjects will receive either Dose level 6 of PMG1015 or Placebo
  Interventions: Drug: PMG1015 Dose 6; Drug: Placebo
- Single Ascending Doses Cohort 1g (Experimental): Subjects will receive either Dose level 7 of PMG1015 or Placebo
  Interventions: Drug: Placebo; Drug: PMG1015 Dose 7

INTERVENTIONS:
Drug: PMG1015 Dose 1 — Dose level 1 of PMG1015
  Other Names: PMG1015
  Arms: Single Ascending Doses Cohort 1a
Drug: PMG1015 Dose 2 — Dose level 2 of PMG1015
  Other Names: PMG1015
  Arms: Single Ascending Doses Cohort 1b
Drug: PMG1015 Dose 3 — Dose level 3 of PMG1015
  Other Names: PMG1015
  Arms: Single Ascending Doses Cohort 1c
Drug: PMG1015 Dose 4 — Dose level 4 of PMG1015
  Other Names: PMG1015
  Arms: Single Ascending Doses Cohort 1d
Drug: PMG1015 Dose 5 — Dose level 5 of PMG1015
  Other Names: PMG1015
  Arms: Single Ascending Doses Cohort 1e
Drug: PMG1015 Dose 6 — Dose level 6 of PMG1015
  Other Names: PMG1015
  Arms: Single Ascending Doses Cohort 1f
Drug: Placebo — Placebo to match
Drug: PMG1015 Dose 7 — Dose level 7 of PMG1015
  Other Names: PMG1015
  Arms: Single Ascending Doses Cohort 1g

SUMMARY:
This is a Phase 1A, first in human, randomized, double-blinded, placebo-controlled, dose escalation study of PMG1015 in healthy adult volunteers. PMG1015 is a monoclonal antibody, being developed as a novel therapeutic treatment for patients with Idiopathic Pulmonary fibrosis (IPF). This study aims to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of PMG1015 after Single ascending doses (SAD).

DETAILED DESCRIPTION:
Participants will be enrolled and randomized into 1 of 7 cohorts in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant, non-lactating female volunteers, between 18 and 60 years of age, inclusive at the time of informed consent.
2. Body mass index (BMI) between 17.5 and 32.0 kg/m2 (inclusive) and body weight between 50 and 100 kg for males and between 45 and 100 kg for females.
3. No clinically significant clinical laboratory values (Hematology, coagulation, biochemistry and urinalysis) at the discretion of the PI.
4. Females of child bearing potential must use an acceptable, highly effective double contraception and have a negative pregnancy test at Screening and Day-1.
5. Documented evidence of surgical sterilization at least 6 months prior to screening for women or vasectomy at least 90 days prior to screening.
6. Women not of child bearing potential must be menopausal for >/= 12 months.
7. Males must not donate sperms for at least 90 days after PMG1015 administration.

Exclusion Criteria:

1. History or evidence of clinically significant condition, including but not limited to any cardiovascular, gastrointestinal, endocrinologic, hematologic, psychiatric, renal disease, musculoskeletal, infectious, or neurological condition or any chronic medical condition and/or other major disease, as determined by the PI.
2. A PR < 40 or > 100 beats per minute, mean systolic blood pressure (SBP) > 140 mmHg, or mean diastolic blood pressure (DBP) > 95 mmHg .
3. A mean corrected QT interval using Fridericia's formula (QTcF) interval at Screening > 450 ms in males and > 470 ms in females. If the mean QTcF exceeds these limits, one additional triplicate ECG will be performed.
4. Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgment of the PI, may interfere with the interpretation of QTc-interval changes, including abnormal ST-T wave morphology or left ventricular hypertrophy.
5. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or creatinine > 1.5 × the upper limit of the normal range (ULN) or total bilirubin or lymphocyte counts > ULN.
6. Participants with a positive toxicology screening panel or alcohol breath test on Screening/Day-1.
7. Participants with a history of substance abuse or dependency or history of recreational IV drug use over the last 2 years.
8. Plasma donation/Blood donation or significant blood loss within 60 days prior to the first IP administration.
9. Use of any IP (including other investigational mAb products) or investigational medical device within 30 days prior to Screening or 5 half-lives of the product (whichever is the longest) or participation in more than 4 investigational drug studies within 1 year prior to screening.
10. Major surgery (general anesthetic) within 3 months or minor surgery (local anesthetic) within 1 month prior to IP administration, or planned surgery during the study period, which is determined by the PI to be clinically relevant.
11. Fever or symptomatic bacterial or viral infection.
12. Participants who have received live vaccines or attenuated vaccines within 1 month before dosing.
13. Participants with any active malignancy or history of malignancy within 5 years prior to enrolment.
14. Use of any other prescription medications.
15. History of anaphylaxis, allergic reactions to the excipients of IP, asthma.
16. Positive blood screen for HIV1/2 antibody, Hepatitis B surface antigen, hepatitis C virus, or syphilis at screening.
17. Participants with an inability to tolerate venous access.
18. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
19. An employee of Pulmongene or Novotech (Australia) Pty Ltd.
20. Participant is unwilling to abstain from alcohol beginning 48 hours prior to admission to the CRU and while resident at the CRU.
21. Any other condition or finding that in the opinion of the PI or designee would put the participant or study conduct at risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
The incidence of Treatment-emergent adverse events (TEAEs) | Day 1-Day 85
  An Adverse Event (AE) is any event, side-effect or any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAEs are AEs that occur following the start of treatment.
The severity of Treatment-emergent adverse events (TEAEs) | Day 1-Day 85
  TEAEs are AEs that occur following the start of treatment.
The incidence of Serious adverse events (SAEs) | Day 1-Day 85
  A serious adverse event (SAE) is defined as an AE occurring during any study phase and at any dose of IP (active or placebo) that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
The severity of Serious adverse events (SAEs) | Day 1- Day 85
  A serious adverse event (SAE) is defined as an AE occurring during any study phase and at any dose of IP (active or placebo) that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
Number of participants with abnormally clinical vital signs | Day 1- Day 85
  Vital signs include pulse rate (PR), blood pressure (BP), respiratory rate (RR) and tympanic temperature (T)
Number of participants with abnormal clinically significant 12-lead electrocardiogram (ECG) parameters | Day 1-Day 85.
  All ECG tracings will be reviewed by the PI or designee and assessed for clinical significance.
Number of participants with abnormal clinically significant clinical laboratory results | Day 1- Day 85
  Clinical laboratory test include hematology, coagulation, biochemistry, and urinalysis.
MTD of PMG1015 in healthy participants | Day 1- Day 85
  Maximum tolerated dose of PMG1015 in healthy participants
Number of patients with abnormal clinically significant results from physical examination | Day 1-Day 85
  Complete physical examination include, general appearance, head, eyes, ears, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.

SECONDARY OUTCOMES:
Area under the serum-concentration time curve (AUC) from time zero (from the start of infusion time) to the last time point with measurable analyte concentration (AUC0-t) | Day 1-Day 85.
  Area under the plasma concentration versus time curve (AUC) from time 0 to time of last quantifiable concentration
AUC from time zero to infinity (AUC0-∞) | Day 1-Day 85.
  Area under the plasma concentration versus time curve (AUC) from time 0 (from the start of infusion) extrapolated to infinity
To determine %AUCexp | Day 1-Day 85.
  The percentage of the AUC that has been extrapolated beyond the last observed data point
To determine Cmax | Day 1-Day 85.
  Maximum observed serum PMG1015 concentration
To determine Tmax, derived from serum concentration of each dose of PMG1015 | Day 1-Day 85.
  Time to maximum observed concentration
To determine t1/2 | Day 1-Day 85.
  Terminal elimination half life summarized by dosing regimen
Apparent total body clearance (CL) | Day 1-Day 85.
  CL is the measure of the rate at which a drug is metabolized or eliminated by normal biological processes
Apparent volume of distribution during the terminal phase (Vz) | Day 1-Day 85.
  Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Apparent terminal elimination rate constant (λz or kel) | Day 1-Day 85.
  λz is calculated using log-linear regression of the terminal portions of the plasma concentrations versus time curves.
Levels of ADA | Day 1-Day 85
  Anti-drug antibody levels in blood

CONTACTS AND LOCATIONS:
Overall Officials: Richard Friend, Principal Investigator — Nucleus Network
Locations (1):
- Q-Pharm Pty Ltd, Clive Berghofer Cancer Research Centre, Herston, Queensland, Australia